CLINICAL TRIAL: NCT02148250
Title: Duration of Action and Peak Effect of High Dose of U-500 Regular Insulin In Severly Insulin Resistant Subjects With Type 2 Diabetes Mellitus
Brief Title: PK/PD Study of U-500 Regular Insulin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1404M49843
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes; Insulin Resistance; High Insulin Requirements
Keywords: Type 2 diabetes; Insulin resistance; High insulin requirements; U 500
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100 Syringe Units, then 200 (Experimental): Participants randomized to first receive 100 syringe units of U-500 regular insulin, then 200 units
  Interventions: Drug: U-500 insulin, 100 syringe units; Drug: U-500 insulin, 200 syringe units
- 200 Syringe Units, then 100 (Experimental): Participants randomized to first receive 200 syringe units of U-500 regular insulin, then 100 units
  Interventions: Drug: U-500 insulin, 100 syringe units; Drug: U-500 insulin, 200 syringe units

INTERVENTIONS:
Drug: U-500 insulin, 100 syringe units — Subjects are randomized to receive 100 syringe units of U-500 insulin. Subjects will receive opposite treatment after 4-8 weeks.
  Other Names: Highly concentrated regular insulin
Drug: U-500 insulin, 200 syringe units — Subjects are randomized to receive 200 syringe units of U-500 insulin. Subjects will receive opposite treatment after 4-8 weeks.
  Other Names: Highly concentrated regular insulin

SUMMARY:
The purpose of this study is to learn more about how U500 regular insulin can be effectively be used to treat type 2 diabetes. Most insulin treated patients with type 2 diabetes take U100 insulin, but if they require large doses (such as >150 units a day) they may experience pain at this site of injection and the absorption of the insulin is unpredictable, thereby leading to poor glucose control. To overcome these problems, doctors sometimes switch to a more concentrated form of insulin called U500 insulin. U500 is five times as concentrated as U100 insulin and therefore delivers an equivalent dose of insulin in much lesser volume. However, how to best use U-500 insulin is not certain. The investigators are not really sure how long a given dose is effective in patients who require large doses (>150 units of U100 insulin), so are not sure of how often the drug should be administered. In this study, the investigators will determine how effective two different doses of U-500 regular insulin (100 U and 200 U) are in lowering blood sugar and how long these two doses last. This information will help doctors develop better treatment plans for patients with type 2 diabetes.

DETAILED DESCRIPTION:
How the Study is performed:

If you agree to participate, you will be given the chance to come to the Masonic Clinical Research Unit (MCRU) at the University of Minnesota for a tour of the facility in the days before the actual experiment. While at the MCRU, one of the investigators will talk with you about the study and provide you with information about the experiments.

During the week before the study, you will be asked to hold oral or injectable non-insulin medicines used to treat diabetes for 1 week prior to the study and to avoid exercise 48 hours prior to the study. During this time you will be asked to monitor your blood sugars and call the investigators for help in managing your sugars if they go outside of the target recommended by your doctor.

On night before the study starts, you will be asked to come to Masonic Clinical Research Unit (MCRU) after dinner (between 8-10 PM). Upon your arrival two catheters will be placed in the arms to establish intravenous access. One will be used for subsequent blood sampling and the other will be used for infusion. We will administer intravenous insulin as necessary to maintain blood glucose between 100-150 mg/dL overnight. Blood sugars will be obtained every 15-60 minutes overnight to ensure the glucose remains at target. At 7 AM the next morning, the intravenous insulin will be stopped. The study will the start when by giving you a dose of either 100 or 200 units of U-500 regular insulin subcutaneously in random order (like a flip of a coin). Since insulin drops the blood sugar, we will also be ready to start an intravenous infusion of glucose to maintain your blood sugars at 100 mg/dl. To keep your sugar at this target, blood will be collected every 15-60 minutes to measure blood sugar and the information will be used by the investigators to figure out how much glucose to give you. We will continue to measure blood glucose until you can maintain blood glucose without a glucose infusion for at least 10 hours or start to experience hyperglycemia (BG > 150 mg/dl) for two hours after discontinuation of the glucose infusion. At that point, the catheters will be removed and you will be discharged to home. During your stay at the MCRU, carbohydrate free meals will be provided starting at noon and continued at traditional mealtimes thereafter for the duration of the glucose infusion. Non-caloric decaffeinated beverages will be available as needed. At the completion of the study you will be told to resume your usual diabetes medications.

Two to four weeks later, you will be asked to once again hold oral or injectable non-insulin medicines used to treat diabetes for 1 week prior to the second part of the study and to avoid exercise 48 hours prior to the study. During this time you will be again asked to monitor your blood sugars and call the investigators for help in managing your sugars if they go outside of the target recommended by your doctor. On night before the second part of the study starts, you will be asked to come to Masonic Clinical Research Unit (MCRU) after dinner. Intravenous lines will again be placed, intravenous insulin will again be given overnight to keep your blood sugar between 100-150 mg/dl, and in the morning you will be given the dose of U500 regular insulin you did not receive during the first visit. Your blood sugar will then be maintained at 100 mg/dl by the infusion of glucose. We will continue to measure blood glucose every 15-60 minutes until you can maintain blood glucose without a glucose infusion for at least 10 hours or start to experience hyperglycemia (BG > 150 mg/dl) for two hours after discontinuation of the glucose infusion. You will be fed the same diet as during your first visit and will be told to resume your diabetes medications at the time we send you home.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Ages 30-65 years
* A1c between 7-9.5% within the past month
* On >100 units of insulin per day
* Willing to discontinue oral/injectable non-insulin hypoglycemic agents for minimum of 1 week prior to study
* Willing to avoid exercise 48 hours prior to study
* Willing to be fasting for up to 24 hours
* BMI between 25 and 38 kg/m2

Exclusion Criteria:

* • On systemic corticosteroids in preceding 3 months

  * Heavy alcohol consumption (>21 drinks/week men, >14 drinks/week women)
  * Unwillingness to stop alcohol consumption for 24 hours before each study visit
  * Pregnant or actively trying to conceive
  * Current diagnosis of active infection, cancer (other than basal cell carcinoma), vascular disease, organ failure
  * Current transplant recipient

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Seaquist, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 100 Syringe Units, Then 200: Participants in this arm were randomized to receive the 100 syringe units of U-500 insulin intervention first, then 200 units.
- 200 Syringe Units, Then 100: Participants in this arm were randomized to receive the 200 syringe units of U-500 insulin intervention first, then 100 units.
Period: Screening
Arm/Group | 100 Syringe Units, Then 200 | 200 Syringe Units, Then 100
Started | 17 | 0
Completed | 12 | 0
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 5 | 0
Period: Period 1
Arm/Group | 100 Syringe Units, Then 200 | 200 Syringe Units, Then 100
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Period 2
Arm/Group | 100 Syringe Units, Then 200 | 200 Syringe Units, Then 100
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: 100 or 200 syringe units of U-500 regular insulin
  U-500 insulin: Subjects are randomized to receive 100 or 200 syringe units of U-500 insulin. Subjects will receive opposite treatment after 4-8 weeks.
Arm/Group | All Subjects
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Duration (in Hours) of 20 % Dextrose Infusion Requirement
Time Frame: 24 hours post insulin injection
Measure: Mean (Standard Deviation); unit: hours
Groups:
- 100 Syringe Units: Arm: 100 syringe units of U-500 regular insulin
- 200 Syringe Units: Arm: 200 syringe units of U-500 regular insulin
Arm/Group | 100 Syringe Units | 200 Syringe Units
Number analyzed (Participants) | 12 | 12
hours | 11 (5.6) | 16.5 (6.4)

2. Secondary Outcome: Peak Infusion Rate Achieved After U-500
Time Frame: 4 hours after insulin injection
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | 100 Syringe Units | 200 Syringe Units
Number analyzed (Participants) | 12 | 12
mg/kg/min | 5.3 (3.8) | 4.2 (1.9)

3. Secondary Outcome: Total Glucose Given After U-500 Dose
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: mg/kg
Groups:
- 200 Syringe Units: Arm: 100 syringe units of U-500 regular insulin
Arm/Group | 100 Syringe Units | 200 Syringe Units
Number analyzed (Participants) | 12 | 12
mg/kg | 5.3 (6.5) | 4.7 (5.6)

4. Secondary Outcome: Time Following Injection the Glucose Infusion Was Started to Maintain EU
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 100 Syringe Units | 200 Syringe Units
Number analyzed (Participants) | 12 | 12
hours | 2.6 (1.3) | 2.2 (1)

5. Secondary Outcome: Total Glucose Required to Maintain Euglycaemia
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | 100 Syringe Units | 200 Syringe Units
Number analyzed (Participants) | 12 | 12
mg/kg | 18.5 (20.7) | 20.1 (13.3)

ADVERSE EVENTS:
Time Frame: Approximately 3 weeks
Arm/Group | 100 Syringe Units | 200 Syringe Units
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT02148250/Prot_SAP_000.pdf